CLINICAL TRIAL: NCT02138175
Title: Continuous Hemoglobin Monitoring: Detection of Acute Blood Loss - Accurate, Timely and Cost-effective
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor (Masimo) suspended trial due to change in corporate ownership
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 03-14-02E
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2015-02

CONDITIONS: Bleeding; Acute Blood Loss Anemia
Keywords: bleeding; blood loss; hemoglobin; hemoglobin monitoring; noninvasive monitoring
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients at risk for bleeding: Patients at risk for bleeding

SUMMARY:
The purpose of the study is to determine whether noninvasive hemoglobin monitoring is sensitive and accurate enough to detect a significant downward trend in hemoglobin in patients at risk for significant bleeding. If this can be shown, it has the potential to spare patients multiple invasive blood draws as well as allow for earlier detection of significant blood loss and therefore positively impact on patient morbidity and mortality. Additionally, it may represent significant financial cost savings in that it may allow for patients to be monitored in a non-intensive care unit setting.

This will be an observational study. The continuous hemoglobin monitor will be connected to the patient and hemoglobin measurement data will be collected. Routine laboratory hemoglobin monitoring will occur concurrently at a pre-specified frequency as well as at the physician's discretion based on usual clinical information. The physician will be blinded to the continuous hemoglobin monitoring readings and therefore patient care will not be affected by the use of the monitor. Once the study has ended, the data will then be analyzed to assess for correlation between continuous hemoglobin monitoring readings and laboratory hemoglobin measurement.

DETAILED DESCRIPTION:
No recruitment initiated

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* admission to surgical intensive care unit
* suspected or high risk for ongoing blood loss

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years) patients admitted to the surgical intensive care unit for hemodynamic monitoring and serial hemoglobin measurements at high risk for bleeding (known solid organ/vascular/orthopedic injury, unexplained hypotension/tachycardia following trauma/surgery, suspected ongoing blood loss-postoperative or gastrointestinal bleeding)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of hemoglobin level measurement between continuous hemoglobin monitor and laboratory analysis | minimum of every 6 hours after intensive care unit admission, shorter intervals if determined indicated by physician based on clinical information, over an estimated period of 3 days, or until patient transferred out of intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Toan Huynh, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Frasca D, Dahyot-Fizelier C, Catherine K, Levrat Q, Debaene B, Mimoz O. Accuracy of a continuous noninvasive hemoglobin monitor in intensive care unit patients. Crit Care Med. 2011 Oct;39(10):2277-82. doi: 10.1097/CCM.0b013e3182227e2d. PMID 21666449
- [Background] Causey MW, Miller S, Foster A, Beekley A, Zenger D, Martin M. Validation of noninvasive hemoglobin measurements using the Masimo Radical-7 SpHb Station. Am J Surg. 2011 May;201(5):592-8. doi: 10.1016/j.amjsurg.2011.01.020. PMID 21545905
- [Background] Coquin J, Dewitte A, Manach YL, Caujolle M, Joannes-Boyau O, Fleureau C, Janvier G, Ouattara A. Precision of noninvasive hemoglobin-level measurement by pulse co-oximetry in patients admitted to intensive care units for severe gastrointestinal bleeds. Crit Care Med. 2012 Sep;40(9):2576-82. doi: 10.1097/CCM.0b013e318258fb4f. PMID 22732278